CLINICAL TRIAL: NCT07230574
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study on Autologous Decidual-like NK Cells Therapy for Reproductive Failure Associated With Abnormal Uterine Natural Killer Cells
Brief Title: Autologous Decidual-like Natural Killer Cells Therapy for Reproductive Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The University of Science and Technology of China (Other); Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Yali Hu, M.D., Ph.D., The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC2025-0013-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Abortion, Missed; Infertility Unexplained; Reproductive Disorder
Keywords: Recurrent Pregnancy Loss; Repeated Implantation Failure; Unexplained Infertility; Decidual Natural Killer Cells
MeSH Terms: conditions — Abortion, Missed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NK cell perfusion group (Experimental): Accepting NK cell therapy
  Interventions: Biological: NK cell perfusion group
- Control group (No Intervention): Not accepting NK cell therapy

INTERVENTIONS:
Biological: NK cell perfusion group — Completing two rounds of NK cell therapy
  Arms: NK cell perfusion group

SUMMARY:
The aim of this study is to verify the efficacy of in vitro induction of autologous decidual-like NK cells therapy for reproductive failure associated with uterine NK cells abnormalities.

DETAILED DESCRIPTION:
Participants with reproductive failure and reproductive intentions will be recruited and screened. After obtaining their informed consent, menstrual blood analysis will be performed. Participants with menstrual blood NK cell abnormalities will be randomly assigned to either the NK cell perfusion group or control group in a ratio of 2:1. After completing two rounds of NK cell therapy, the NK cell perfusion group will enter the follow-up period, while the control group will not receive interventions after randomization and enter the follow-up period directly. The following information will be recorded for all participants who undergo menstrual blood NK cell analysis, including menstrual blood analysis results, attempts to conceive, and pregnancy outcomes during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive failure with abnormal endometrial natural killer (NK) cells in menstrual blood;
* With a clear intention to conceive;
* Normal ovarian function, or premature ovarian insufficiency with ≥2 high-quality cryopreserved embryos available for transfer;
* Endometrial thickness measured by transvaginal ultrasound during the periovulatory period ≥7 mm;
* Body mass index (BMI) between 18 kg/m² and 28 kg/m²;
* Willing to comply with the follow-up plan of this study.

Exclusion Criteria:

* Use of progesterone receptor modulators;
* One of the couple's chromosomal karyotype abnormalities, with no euploid embryo identified via preimplantation genetic testing for aneuploidy;
* Severe endometriosis or adenomyosis, uterine fibroids affecting uterine cavity morphology, uterine malformations, intrauterine adhesions, or thin endometrium;
* Uncontrolled autoimmune or endocrine disorders;
* Contraindications to pregnancy;
* History of malignant tumors;
* Participating in other clinical studies;
* Allergy to blood products.

Ages: 22 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 6 months, if a participant is confirmed to get a clinically pregnancy during this period, the follow-up endpoint will be extended until there is a pregnancy outcome
  Ongoing pregnancy is defined as at least 12 weeks of gestation, with ultrasound indicating fetal cardiac activity and fetal size consistent with the gestational age

SECONDARY OUTCOMES:
Improvement rate of NK cells | 6 months
  Improvement rate of NK cells in menstrual blood analysis after intrauterine perfusion of autologous decidual-like NK cells
Clinical pregnancy rate | 6 months
  Clinical pregnancy is defined as the presence of a gestational sac in the uterine cavity as indicated by ultrasound at 5-7 weeks of gestation
Miscarriage rate | 6 months, if a participant is confirmed to get a clinically pregnancy during this period, the follow-up endpoint will be extended until there is a pregnancy outcome
  Miscarriage is defined as the pregnancy loss before 28 weeks of gestation
Preterm birth rate | 6 months, if a participant is confirmed to get a clinically pregnancy during this period, the follow-up endpoint will be extended until there is a pregnancy outcome
  Preterm birth is defined as delivery at 28 to 37 weeks of gestation
Live birth rate | 6 months, if a participant is confirmed to get a clinically pregnancy during this period, the follow-up endpoint will be extended until there is a pregnancy outcome
  Live birth is defined as delivery of any number of neonates born at 26 or more weeks' gestation with signs of life

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University